CLINICAL TRIAL: NCT00648726
Title: An Open, Prospective, Randomized, Multi-Center Study of the Efficacy and Safety of Intravenous Followed by Oral Azithromycin vs. Cefuroxime Monotherapy or Plus Oral Erythromycin for the Treatment of Chinese Hospitalized Patients With Community- Acquired Pneumonia
Brief Title: An Open, Prospective, Randomized, Multicenter Study of the Efficacy and Safety of Intravenous Followed by Oral Azithromycin Versus Cefuroxime Alone or With Oral Erythromycin for the Treatment of Chinese Patients Who Were Hospitalized for Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0661104
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Cefuroxime; Erythromycin; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: cefuroxime plus erythromycin
- Arm 2 (Active Comparator)
  Interventions: Drug: azithromycin (Zithromax)
- Arm 3 (Active Comparator)
  Interventions: Drug: cefuroxime

INTERVENTIONS:
Drug: cefuroxime plus erythromycin — intravenous cefuroxime 1.5 g twice daily for 4 +/-1 days, followed by oral cefuroxime 0.5 g twice daily for a total duration of 9 +/-1 days plus erythromycin ethylsuccinate 0.5 g twice daily, which was given for a total duration of 14 days for subjects with suspected pneumonia due to atypical pathogens
  Arms: Arm 1
Drug: azithromycin (Zithromax) — intravenous azithromycin 500 mg once daily for 4 +/-1 days, followed by oral azithromycin 500 mg once daily for a total duration of 9 +/-1 days
  Arms: Arm 2
Drug: cefuroxime — intravenous cefuroxime 1.5 g twice daily for 4 +/-1 days, followed by oral cefuroxime 0.5 g twice daily for a total duration of 9 +/-1 days
  Arms: Arm 3

SUMMARY:
To validate the efficacy and safety of azithromycin for the treatment of Chinese patients hospitalized with community-acquired pneumonia (CAP), compared with cefuroxime or the combination of cefuroxime plus oral erythromycin.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Patients hospitalized with a diagnosis of community acquired pneumonia (CAP) as defined by the presence of new infiltrate(s) including manifestation of consolidation, patchy, diffuse or interstitial inflammation on chest X-ray with or without pleural effusion plus at least 1 of the following: new cough and expectoration or progression of respiratory symptoms with purulent sputum with or without chest pain; fever; auscultatory findings such as rales or evidence of pulmonary consolidation; blood leukocyte count >10×109/L or <4×109/L with or without >15% bands or a blood leukocyte count between 4 and 10 with neutropils greater than or equal to 75%

Exclusion Criteria:

Exclusion Criteria:

* Patients with hospital acquired pneumonia, aspiration pneumonia, severe pneumonia, history of post-obstructive pneumonia, active tuberculosis or bronchitis, bronchiectasis or chronic obstructive pulmonary disease without evidence of acute infection were not eligible for this study
* Patients treated with any systemic antibiotic within 72 hours prior to study entry were not eligible unless the medication was, in the opinion of the investigators, classified as having failed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2003-01; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
clinical efficacy (cure or marked improvement) | Visit 3 (Day 9 +-1 of treatment)

SECONDARY OUTCOMES:
bacteriological efficacy (eradication) | Visit 3
clinical efficacy | Visit 4 (8 +/-1 days after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661104&StudyName=An%20Open%2C%20Prospective%2C%20Randomized%2C%20Multicenter%20Study%20of%20the%20Efficacy%20and%20Safety%20of%20Intravenous%20Followed%20by%20Oral%20Azithromycin%20Versus%20C